CLINICAL TRIAL: NCT00362557
Title: Body Magnetic Resonance (MR) Imaging Techniques
Brief Title: Imaging Techniques in Body Magnetic Resonance Imaging "MRI"
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00067074
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Clinically Indicated MR Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: MRI — Magnetic resonance imaging

SUMMARY:
Any patient already receiving a scheduled MR scan of the body for any clinical indication will be eligible for this program.

DETAILED DESCRIPTION:
If patients agree to participate in this program, it would require only a slightly longer examination time. This time would vary according to the body area/organ being visualized but would not exceed 30 minutes over the length of the clinical examination. Volunteers are eligible if they are willing to undergo an MR examination.

Patients would not be required to make any additional visits beyond their clinically-indicated visits. The study duration would vary according to the body area/organ visualized but would not exceed 30 minutes over the length of the clinical examination. Volunteers would be required to keep one study appointment to include one MR imaging examination.

There will be no interruption to the standard care given to patients who participate in this trial since the clinical portion of their examination will be completed prior to the study portion of the exam.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female clinically scheduled to undergo MR Imaging at Johns Hopkins Medical Institutions

Exclusion Criteria:

* Contraindications to MR Imaging

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who may require a body MRI examination
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2001-09; Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Magnetic resonance signal | One Hour
  Magnetic resonance imaging acquires signal from the human body. The signal will be measured at the time of the patient study. The amount of signal change will be measured between subjects.

CONTACTS AND LOCATIONS:
Overall Officials: David A Bluemke, MD PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Pontiff M, Moreau NG. Safety and Feasibility of 1-Repetition Maximum (1-RM) Testing in Children and Adolescents With Bilateral Spastic Cerebral Palsy. Pediatr Phys Ther. 2022 Oct 1;34(4):472-478. doi: 10.1097/PEP.0000000000000941. Epub 2022 Aug 12. PMID 35960137